CLINICAL TRIAL: NCT06348095
Title: Effect of Probiotic WecProB on the Course of Mycoplasma Pneumoniae Pneumonia in Children
Brief Title: Effect of Probiotics on Mycoplasma Pneumoniae Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2024004
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mycoplasma Pneumoniae Pneumonia
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): 2B CFU/ strip/ day WecProB, before meals; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Maltodextrin, one strip/ day WecProB, before meals; Storage: Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study had last 14 days, and each patient will make 4 visits (d0, d3, d7, d14).
  Arms: Probiotics group
Dietary Supplement: Placebo — The experimental phase of this study had last 14 days, and each patient will make 4 visits (d0, d3, d7, d14).
  Arms: Placebo group

SUMMARY:
To evaluate the effectiveness and safety of compound probiotic in shortening the course of illness in children with mycoplasma pneumoniae pneumonia, in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for pneumonia in "Zhufutang Practical Pediatrics" (7th Edition), and is diagnosed with Mycoplasma pneumoniae pneumonia using tNGS technology;
2. Infants and young children aged 6 months to 3 years;
3. The course of the disease is <48 h;
4. The family members of the children are informed about the study and sign the informed consent form.

Exclusion Criteria:

1. Previous history of wheezing;
2. Cardiovascular disease and congenital tracheal dysplasia;
3. pneumonia induced by other causes;
4. Dysplasia of bronchial and pulmonary tracts;
5. premature infants;
6. Combined with immunosuppressive diseases;
7. Presence of mental illness.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-05-27 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mycoplasma pneumoniae load | 7天
  Mycoplasma pneumoniae load was detected by tNGS